CLINICAL TRIAL: NCT02315391
Title: Efficacy of Isolated Whey and Micellar Whey Protein (+/- Citrulline) to Stimulate Protein Synthesis in 'Healthy' and 'Anabolically Resistant' Elderly Muscle
Brief Title: Protein Nutrition for Muscle Hypertrophy in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11.06.NRC
Record Dates: First submitted 2014-11-12; First posted 2014-12-11 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Elderly Muscle; Anabolically Resistant Elderly Muscle
MeSH Terms: interventions — Glycine; Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20g isolated whey protein + 30g carb, 8,5g fat, 15g glycine (Experimental): 20g isolated whey protein + 30g carb, 8,5g fat, 15g glycine
  Interventions: Dietary Supplement: isolated whey protein; Dietary Supplement: glycine
- 20g micellar whey protein + 30g carb, 8.5g fat, 15g glycine (Experimental): 20g micellar whey protein + 30g carb, 8.5g fat, 15g glycine
  Interventions: Dietary Supplement: micellar whey protein; Dietary Supplement: glycine
- 20g micellar whey protein + 30g carb, 8.5g fat, 5g citrulline (Experimental): 20g micellar whey protein + 30g carb, 8.5g fat, 5g citrulline
  Interventions: Dietary Supplement: micellar whey protein; Dietary Supplement: citrulline

INTERVENTIONS:
Dietary Supplement: isolated whey protein — isolated whey protein
  Arms: 20g isolated whey protein + 30g carb, 8,5g fat, 15g glycine
Dietary Supplement: micellar whey protein — micellar whey protein
  Arms: 20g micellar whey protein + 30g carb, 8.5g fat, 15g glycine; 20g micellar whey protein + 30g carb, 8.5g fat, 5g citrulline
Dietary Supplement: glycine — glycine
  Arms: 20g isolated whey protein + 30g carb, 8,5g fat, 15g glycine; 20g micellar whey protein + 30g carb, 8.5g fat, 15g glycine
Dietary Supplement: citrulline — citrulline
  Arms: 20g micellar whey protein + 30g carb, 8.5g fat, 5g citrulline

SUMMARY:
The primary objective is to determine the effect of reduced activity on the stimulation of myofibrillar FSR with protein feeding in the elderly.

DETAILED DESCRIPTION:
The primary objective is to determine the effect of reduced activity on the stimulation of myofibrillar FSR with protein feeding in the elderly

ELIGIBILITY:
Inclusion Criteria:

* Must habitually complete a minimum of 5000 steps per day
* Having obtained informed consent
* Non-obese
* Non-smoker

Exclusion Criteria:

* Aged >80 years
* Inability to comply with study procedures
* Currently participating or having participated in another infusion trial during last 12 months
* Any acute or chronic llness
* History of neuromuscular problems
* Medications known to affect protein metabolism
* Individuals who complete fewer than 5000 steps per day
* Individuals who have metal implants

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in myofibrillar fractional synthetic rate (FSR) | one day and 2 weeks

SECONDARY OUTCOMES:
change in non-myofibrillar fractional synthetic rate (FSR) | baseline and one day of feeding
Capillary dilatation and blood flow | 2 weeks
  Determine if inactivity reduces the feeding-induced increase in capillary dilation and nutrient delivery and whether citrulline rescues this in "resistant" muscle or augments it in the "healthy" muscle as measured by Definity infusion and contrast enhanced ultrasound (CEUS)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Philips, PhD, Principal Investigator — McMaster University